CLINICAL TRIAL: NCT00006144
Title: A Phase II Exploratory Study Examining Immunologic and Virologic Indices in Two Age-Differentiated Cohorts of HIV-Infected Subjects to Explore the Basis of Accelerated HIV-Disease Progression Associated With Aging
Brief Title: A Study of HIV-Disease Development in Aging
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: A5015; 10168 (Registry Identifier: DAIDS ES); ACTG A5015; AACTG A5015; Substudy ACTG A5016s; Substudy ACTG A5020s
Record Dates: First submitted 2000-08-07; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Stavudine; HIV Protease Inhibitors; Cohort Studies; Ritonavir; Disease Progression; Antigens, CD; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Immunophenotyping; Deoxycytidine
MeSH Terms: conditions — HIV Infections; Disease Progression | interventions — Lopinavir; Emtricitabine; Stavudine

INTERVENTIONS:
Drug: Lopinavir/Ritonavir
Drug: Emtricitabine
Drug: Stavudine

SUMMARY:
The purpose of this study is to better understand the relationship between age and HIV disease progression.

This study will explore the possible relationship between age and HIV disease progression. Older age is an important risk factor for faster disease development, but older people may respond better to combination drug therapy. This relationship needs to be understood better.

DETAILED DESCRIPTION:
Older age is an important risk factor for accelerated HIV-disease progression. However, the virologic response to highly active antiretroviral therapy (HAART) may be superior in older persons. A better understanding of the immunologic, virologic, and behavioral mechanisms that underlie these age-related differences may help to elucidate critical immune responses that are necessary to control the progression of HIV-disease.

Patients are grouped according to age. Group A consists of patients between the ages of 13 and 30 years. Group B consists of patients age 45 years or older. All patients receive open-label lopinavir/ritonavir (LPV/RTV) plus emtricitabine (FTC) plus stavudine (d4T) for 96 [AS PER AMENDMENT 06/04/02: 192] weeks. Study visits occur at pre-entry, entry, and Weeks 4, 8, 12, 16, and 24 then every 12 weeks thereafter through Week 96 [AS PER AMENDMENT 06/04/02: Week 192]. Clinical assessments, safety laboratory tests, CD4 cell count monitoring, lymphocyte phenotyping, and HIV-1 RNA determinations are performed routinely. Blood samples are stored for further immunology and virology studies. Patients may volunteer to participate in virology substudy A5020s and either immunology substudy A5016s or A5017s [AS PER AMENDMENT 06/04/02: Substudy A5017s has been eliminated.]

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Are between 13 and 30 years old (need consent of parent or guardian if under 18), or are more than 44 years of age.
* Have a viral load of more than 2000 copies/ml within 60 days of study entry.
* Have a CD4 cell count of less than 600 cells/mm3 within 60 days of study entry. (This reflects a change in the CD4 cell count requirement.)
* Agree to use effective methods of birth control (such as condoms) during and for 12 weeks after the study.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Are pregnant or breast-feeding.
* Have an AIDS-related cancer (except Kaposi's sarcoma) requiring chemotherapy.
* Have hepatitis within 30 days of study entry.
* Have diarrhea (more than 3 liquid stools/day for at least 14 days) within 30 days of study entry.
* Are receiving chemotherapy or radiation treatment.
* Have taken antiretroviral drugs for more than 14 days.
* Have received an HIV vaccine within 30 days of study.
* Have a serious illness or infection within 14 days of the study.
* Have other serious conditions that might interfere with study participation.
* Have taken or plan to take certain other drugs that might affect the study results.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90
Dates: Start 2000-10; Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kalayjian, Study Chair; Michael Lederman, Study Chair; Richard Pollard, Study Chair
Locations (45):
- United States (44):
  - USC CRS, Los Angeles, California
  - Stanford CRS, Palo Alto, California
  - Ucsf Aids Crs, San Francisco, California
  - Santa Clara Valley Med. Ctr., San Jose, California
  - San Mateo County AIDS Program, San Mateo, California
  - Marin County Dept. of Health & Human Services, HIV/AIDS Program & Specialty Clinic, San Rafael, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Queens Med. Ctr., Honolulu, Hawaii
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Northwestern University CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Indiana Univ. School of Medicine, Wishard Memorial, Indianapolis, Indiana
  - Methodist Hosp. of Indiana, Indianapolis, Indiana
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Bmc Actg Crs, Boston, Massachusetts
  - Brigham and Women's Hosp. ACTG CRS, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - SSTAR, Family Healthcare Ctr., Fall River, Massachusetts
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - Washington U CRS, St Louis, Missouri
  - Beth Israel Med. Ctr., ACTU, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Mt. Sinai Med. Ctr. A0404 CRS, New York, New York
  - Columbia Univ., HIV Prevention and Treatment Medical Ctr., New York, New York
  - Mt.Sinai Med. Ctr. A1009 CRS, New York, New York
  - Trillium Health ACTG CRS, Rochester, New York
  - AIDS Care CRS, Rochester, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - Case CRS, Cleveland, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - Philadelphia Veterans Admin. Med. Ctr. A6205 CRS, Philadelphia, Pennsylvania
  - The Miriam Hosp. ACTG CRS, Providence, Rhode Island
  - Rhode Island Hosp., Providence, Rhode Island
  - Vanderbilt Therapeutics CRS, Nashville, Tennessee
  - Univ. of Texas Southwestern Med. Ctr., Amelia Court Continuity Clinic, Dallas, Texas
  - Univ. of Texas Medical Branch, ACTU, Galveston, Texas
  - University of Washington AIDS CRS, Seattle, Washington
- Puerto Rico-AIDS CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Kalayjian R, Landay A, Pollard R, Pu M, Spritzer J, Tebas P, Gross B, Valcour V, Cu-Uvin S, Fiscus S, Fidel P, Wu A, Fox L, Stocker V, Lederman M, and AIDS Clinical Trials Group Protocol 5015. ACTG 5015: NaIve T-cell Reconstitution is Associated with Immune Activation. CROI 2004. Abstract 232.
- [Derived] Tenorio AR, Spritzler J, Martinson J, Gichinga CN, Pollard RB, Lederman MM, Kalayjian RC, Landay AL. The effect of aging on T-regulatory cell frequency in HIV infection. Clin Immunol. 2009 Mar;130(3):298-303. doi: 10.1016/j.clim.2008.10.001. Epub 2008 Nov 12. PMID 19008157